CLINICAL TRIAL: NCT00291122
Title: Quantitative Real Time PCR in Formalin Fixed Breast Tissue From Biopsy and Re-Excision Specimens: An Ancillary Protocol to a Chemoprevention Trial of Celecoxib
Brief Title: An Examination of Predictors of Indicators of Response to Celecoxib in Women Who Have a Diagnosis of Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 9380
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: breast atypia; breast epithelial hyperplasia; ki-67; RTPCR; microdissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; BID protein, human

INTERVENTIONS:
Drug: celecoxib 400 mg BID

SUMMARY:
To assess the quantitative real time PCR results results of oligonucleotide probes for a number of gene transcription products that may be useful as predictors of indicators of response to celecoxib.

DETAILED DESCRIPTION:
To assess the quantitative real time PCR results of oligonucleotide probes for a number of gene transcription products that may be useful as predictors or indicators of response to celecoxib, the feasibility of performing six different molecular assays by qRTPCR on formalin fixed paraffin embedded tissue obtained from breast cancer core biopsies and breast cancer reexcision patients, to assess change in Ki-67, PCNA, and several other markers by qRTPCR, correlate change in expression of Ki-67, PCNA, CAX-2, and bcl-2, measured by immunohistochemistry to change measured by qRTPCR, and to determine the reliability of the qRTPCR and immunohistochemical assays by performed selected assays on the same tissue in two different institutions

ELIGIBILITY:
Inclusion Criteria:

* women with a recent diagnosis of T1 or T2 noninvasive breast cancer by large core needle or excisional biopsy
* confirmation that tissue was processed in methods acceptable to protocol and sufficient tissue remains post diagnostic analyses to perform research assessments
* reexcision planned within 10 days to 6 weeks from study start

Exclusion Criteria:

* no hormone replacement therapy within 90 days prior to biopsy
* no history of asthma, allergy ASA, NSAIDS, celecoxib of other COX-2 inhibitors for a chronic non-oncological condition with the excision of low dose ASA (160 mg daily) during 4 weeks prior to biopsy and for the duration of the study
* no celecoxib or rofecoxib use within one month of biopsy
* no history of gastrointestinal ulcer or ulcerative colitis requiring treatment
* no current anticoagulants
* no neoadjuvant antihormone or chemotherapy as treatment following biopsy prior to study entry or concurrently with participation on study
* no aromatase inhibitor in the six months prior to participation
* no concomitant lithium
* no known significant bleeding disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States